CLINICAL TRIAL: NCT04017702
Title: Detection of Postoperative Respiratory Depression in High Risk Patients Utilizing Minute Ventilation Monitoring
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000021197
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Respiratory Depression
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Pregnant women with gestational age between 32-40 weeks.: 100 patients scheduled for cesarean section under neuraxial anesthesia with 150 mcg intrathecal or 3-mg epidural morphine.
- Patients post anesthesia care units (PACU) and surgical floor.: 100 patients scheduled to receive General Anesthesia (GA) and planned to receive opioid intravenously (boluses/patient controlled analgesia (PCA).
- Patients in step down/ICU.: 50 patients suffered from rib fracture and 50 patients after weaning from mechanical ventilation and extubation.The Expiron will provide continuous information about the respiratory status (tidal volume, respiratory rate and minute ventilation) of non-intubated patients specifically: sleeping or awake; with the use of incentive spirometry; the response to medications and other interventions (such as paravertebral/epidural block); the need for endotracheal re-intubation.
  Interventions: Device: Expiron respirator

INTERVENTIONS:
Device: Expiron respirator — Respiratory volume monitor (RVM) (ExSpiron, is a non-invasive FDA approved device that monitors minute ventilation (MV) and provides an early indication of respiratory status in non-intubated patients. The system consists of a lightweight monitor, a patient cable, and a disposable electrode PadSet, which detects changes in breathing.
  Groups: Patients in step down/ICU.

SUMMARY:
Respiratory volume monitor (RVM) (ExSpiron) is superior to continuous pulse oximetry in detection of postoperative respiratory depression in high risk patients.

DETAILED DESCRIPTION:
Aims are to: 1) Estimate the incidence of postoperative respiratory depression in high risk patients as detected by continuous pulse oximetry 2) Estimate the incidence of postoperative respiratory depression in high risk patients as detected by continuous respiratory volume monitor (RVM) (ExSpiron) 3) Assess the agreement between the continuous pulse oximetry and continuous respiratory volume monitor (RVM) (ExSpiron) in detection of postoperative respiratory depression in high risk patients

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffered rib fractures or patients who are weaned from mechanical ventilation and recently extubated.

Exclusion Criteria:

* Have known contraindication/allergy to neuroaxial/paravertebral nerve block anesthesia
* Patients allergic to morphine.
* Have an ASA class > IV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group A; which will involve pregnant women with gestational age between 32-40 weeks. It will take place at:
  i. Labor and delivery floor/obstetric floor: 100 patients scheduled for cesarean section under neuraxial anesthesia with 150 mcg intrathecal or 3-mg epidural morphine.
  ii. Antenatal care: (obstetric floor, Long Wharf women clinic, Women center at Yale)
  Group B; in post anesthesia care units (PACU) and surgical floor: 100 patients scheduled to receive General Anesthesia (GA) and planned to receive opioid intravenously (boluses/patient controlled analgesia (PCA).
  Group C: in step down/ICU; 50 patients suffered from rib fracture and 50 patients after weaning from mechanical ventilation and extubation.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative respiratory depression | 1 year
  To define the incidence of postoperative respiratory depression between 2 devices.

SECONDARY OUTCOMES:
Detection of postoperative respiratory depression in high risk patients. | 1 year
  To determine the agreement between these 2 devices in detection of postoperative respiratory depression in high risk patients.

CONTACTS AND LOCATIONS:
Overall Officials: Aymen Alian, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States